CLINICAL TRIAL: NCT04856943
Title: Evaluation of the Effectiveness of Smartconsent to Improve Understanding of Informed Consent in Prostate Laser Enucleation Procedures
Brief Title: Effectiveness of Smartconsent in Improving Understanding of Informed Consent
Acronym: SMARTCONSENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bioaraba Health Research Institute (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SMARTCONSENT
Record Dates: First submitted 2021-04-20; First posted 2021-04-23 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- smartconsent group (Experimental): Intervention group: : the principal investigator upon receiving the tablet enters with his/her user and password, registers his/her signature, selects the patient (anonymized), selects the intervention and then the tablet will be given to the patient and he/she will be instructed to follow the indications in order to be able to project the video and digitally sign the informed consent.
  Interventions: Procedure: Smartconsent application
- control group (Placebo Comparator): Control group: The informed consent paper document (official format) will be printed with the patient's name, signed by the physician (principal investigator) and given to the patient to read and sign.
  Interventions: Other: Control group

INTERVENTIONS:
Procedure: Smartconsent application — Patients asigned to smartconsent group will sign informed consent through a Tablet.
  Arms: smartconsent group
Other: Control group — Patient asigned to control group will sing the informed consent in papel, as it is performed in clinical practice
  Arms: control group

SUMMARY:
The general objective of the study is to assess whether the new smartconsent tool improves patients' understanding of the intervention to be performed, compared to standard practice.

A randomized clinical trial will be conducted in 50 patients who will undergo LASER PROSTATIC ENUCLEATION.

DETAILED DESCRIPTION:
Male patients aged between 50 and 70 years, belonging to the Hospital Universitario Araba who are going to undergo PROSTATIC LASER ENUCLEATION, and who attend urology consultation between December 2019 and December 2020, and who meet the inclusion criteria and none of the exclusion criteria.

Inclusion criteria:

* Patients willing to receive information via tablet.
* Patients who know how to and can read.

Exclusion criteria:

-Not applicable.

Main variable: score on the Multiple choice test questionnaire (designed specifically for each type of procedure, following the recommendations proposed by Kehoe, Jerard and Fathelrahman et al. and developed on the basis of the information that an informed consent should provide (1, 2), with 4 response options and only one correct answer. An average score will be calculated for each patient.

This test evaluates the comprehension of the information provided through the informed consent.

ELIGIBILITY:
Inclusion criteria:

* Patients willing to receive information via tablet.
* Patients who know and can read.

Exclusion Criteria:

* Not applicable

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2021-12-31 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Score in the Multiple choice test questionnaire | At the recruitment moment
  Specifically designed for each type of procedure, following the recommendations proposed by Kehoe, Jerard and Fathelrahman et al. and developed on the basis of the information to be provided in an informed consent form, with 4 response options and only one correct answer

SECONDARY OUTCOMES:
Satisfaction with the informed consent proccess | At the recruitment moment
  based on three ad hoc designed items: Each item will be scored on a lipo Likert scale with 5 response options.
Ability to complete the informed consent form | At the recruitment moment
  Without the need for additional information from the healthcare professional.
Time required to complete the informed consent process (MIN). | At the recruitment moment
  The Smartphone stopwatch of the researchers participating in the study will be used for this purpose
Overall satisfaction with the informed consent process, | At the recruitment moment
  Through a three-item test, developed ad hoc by a group of researchers to assess satisfaction in a study with similar characteristics to ours.
Score in the System Usability Scale | At the recruitment moment
  In the SMARTCONSENT group only. he average System Usability Scale score is 68. If your score is under 68, then there are probably serious problems with your website usability which you should address. If your score is above 68, then you can relax a little bit.

CONTACTS AND LOCATIONS:
Overall Officials: IMANOL MERINO, Principal Investigator — Bioaraba Health Research Institute
Locations (2):
- Spain (2):
  - Imanol Merino, Vitoria-Gasteiz, Alava
  - Bioaraba Health Research Institute, Vitoria-Gasteiz, Alava